CLINICAL TRIAL: NCT07266519
Title: SIRIUS - A Prospective, Non-randomized, Open-label, Proof-of-concept Study of Initial Combination Therapy With an Endothelin Receptor Antagonist, a Phosphodiesterase-5 Inhibitor and Sotatercept in Patients With Newly Diagnosed Pulmonary Arterial Hypertension A Single-arm, Multi-center, Interventional Phase II Study
Brief Title: SIRIUS - Initial Combination Therapy With an Endothelin Receptor Antagonist, a Phosphodiesterase-5 Inhibitor and Sotatercept in Patients With Newly Diagnosed Pulmonary Arterial Hypertension
Acronym: SIRIUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: MSD Sharp & Dohme GmbH, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KKS-322; 2025-522266-67-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: triple therapy; PAH; treatment-naiive
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized, multi-center, proof-of-concept
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Treatment arm
  Interventions: Drug: Sotatercept 0.3 mg/kg escalating to 0.7 mg/kg; Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept 0.3 mg/kg escalating to 0.7 mg/kg — subcutaneously administration in 3-weekly intervals
Drug: Sotatercept — Patients are traitment-naiive before start of study. Therapy will be a triple combination therapy with an endothelin receptor antagonist (ERA), a phosphodiesterase-5 inhibitor (PDE5i), and Sotatercept

SUMMARY:
The study aims to see how 24 weeks of triple therapy-an endothelin receptor antagonist (ERA), a phosphodiesterase-5 inhibitor (PDE5i), and sotatercept-affects pulmonary vascular resistance (PVR) in patients with newly diagnosed pulmonary arterial hypertension (PAH). SIRIUS is a 24-week, single-arm, open-label study with up to 42 days of screening and a 28-day safety follow-up. It will enroll 25 patients and will be conducted only in countries where all treatments are available and covered. After 24 weeks, PAH treatment is decided by the doctor.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 70 years
* Treatment-naïve patients diagnosed within 12 weeks prior to screening with I/H/D-PAH or PAH associated with corrected congenital heart disease (disease (≥12 months after correction). Patients who have received treatment with PDE5is and/or ERAs for up to 6 weeks after diagnosis are eligible provided that state-of-the-art right heart catheterization has been performed at PAH diagnosis.
* PVR >5 WU, mPAP ≥35 mmHg and PAWP or LVEDP ≤15 mmHg at PAH diagnosis.
* Signed written informed consent
* Normal blood counts for platelets and erythrocytes
* Women of childbearing potential must be willing to remain abstinent or use adequate and reliable contraception throughout the study and for at least 4 months after the last dose of study medication has been received.

  * WOCBP must use one of the following highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly - according to recommendations by the European Heads of Medicines Agencies - from at least 14 days before the first administration of study medication until 4 month after the last administration of study medication:
  * combined (estrogen and progestogen containing) hor-monal contraception associated with inhibition of ovulation:

    * oral
    * intravaginal
    * transdermal
  * progestogen-only hormonal contraception associatedwith inhibition of ovulation:

    * oral
    * injectable
    * implantable
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system (IUS)
  * bilateral tubal occlusion
  * vasectomized partner
  * sexual abstinence
* Male participants with female partner(s) of childbearing potential are eligible to participate in the study if they agree to the following during treatment and until 304 daysmonths after the last administration of study medication:

  * Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
  * Male participants are required to use a condom during treatment and until 30 days4 months after the last administration of study medication.
  * Female partners of male participants who have not undergone a vasectomy with the absence of sperm confirmed or a bilateral orchiectomy should consider use of effective methods of contraception during treatment and until 30 days4 months after the last administration of study medication.
* Sperm donation is not allowed during treatment and until 4 months after the last administration of study medication.

Exclusion Criteria:

* Other Forms of PH or PAH
* Use of PAH medications for more than 6 weeks prior to screening
* Symptoms or signs of clinically relevant lung disease, including TLC < 70%, FEV1/FVC <60%, and DLCO <45%, respectively
* Signs of left heart failure with reduced or preserved ejection fraction, including LVEF <50%, LAVI >34 ml/m2, E/é ≥15, or permanent atrial fibrillation, respectively.
* History of severe bleeding/haemorrhage
* Therapy with prostacyclin and/or antithrombotic agents
* eGFR <30 ml/min/m2.
* Pregnancy or breastfeeding
* Hypersensitivity to the active substance or to any of the excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effect on pulmonary vascular resistance (PVR) | 24 weeks
  Change in PVR from screening at week 24 after 6-months of treatment with triple combination therapy in PAH patients

CONTACTS AND LOCATIONS:
Overall Officials: Karen Olsson, Prof. Dr., Principal Investigator — Hannover Medical School Department of Respiratory Medicine

IPD SHARING:
Plan to Share IPD: Undecided